CLINICAL TRIAL: NCT01552460
Title: Brain Genomics Superstruct Project
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Clinical Investigator, Clinical and Research Program in Pediatric Psychopharmacology and Adult ADHD, Massachusetts General Hospital
Other Study IDs: 2011P000375
Record Dates: First submitted 2012-03-01; First posted 2012-03-13 (Estimated); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorders
Keywords: Autism Spectrum Disorders; Brain Imaging; Genetics
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to explore the effects of genes and genetic variation on brain structure and function. Investigators at Harvard plan to explore the relationship between candidate genes that affect cognitive performance and brain structure/function. Since brain phenotypes reflect more proximal sequelae of gene activity, neuroimaging measures may show greater sensitivity than cognitive performance to measure gene effects.

ELIGIBILITY:
Inclusion Criteria:

1. 13 years or older
2. Subject must have a current DSM-IV diagnosis of high functioning ASD, based on past evaluations at the Bressler Clinic.
3. Subjects must have a level of understanding sufficient to communicate intelligently with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
4. Each subject must understand the nature of the study. The subject must sign an IRB approved informed consent.

Exclusion Criteria:

1. IQ < 70 bassed on evaluation in the Bressler Clinic.
2. Contraindication to MRI including presence of metal or surgical devices (plates, implants, braces or other items).
3. Neuropsychiatric conditions (such as dementia) which sufficiently impair cognition such that a surrogate consent would be required.
4. Neurological disorders associated with gross brain pathology (other than atrophy), e.g., stroke, tumors, or demyelinating diseases.
5. Pregnancy.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults with Autism Spectrum Disorders ages 13 and older.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2011-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Neuroimaging phenotype | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States